CLINICAL TRIAL: NCT02013583
Title: The Glucose Transporter Type I Deficiency (G1D) Registry
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Juan Pascual, Associate Professor, Director of the Rare Brain Disorders Program, University of Texas Southwestern Medical Center
Other Study IDs: UTSW 062012-080
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: GLUT1 Deficiency Syndrome; Glucose Transporter Type 1 Deficiency Syndrome; Glucose Transporter Type1 (GLUT-1) Deficiency; GLUT-1 Deficiency Syndrome
Keywords: Glucose Transporter Type I Deficiency; Glucose Transporter Type 1 Deficiency; G1D; Glut1 Deficiency
MeSH Terms: conditions — Glut1 Deficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glucose Transporter Type I Deficiency: No interventions
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational registry. No interventions are required or provided.

SUMMARY:
The purpose of this protocol is to create a registry for patients diagnosed with Glucose Transporter Type 1 Deficiency (G1D), or patients experiencing symptoms consistent with G1D but not yet diagnosed, to enter medical information for physicians and other health researchers to analyze to increase the understanding of G1D and any sub-diagnoses.

DETAILED DESCRIPTION:
This is a registry for patients diagnosed with G1D, or experiencing symptoms G1D but not yet diagnosed. The registry will be available online for patients to provide consent, register, enter data, and modify data as necessary. The registry will be programmed by programmers at UT Southwestern Medical Center. The registry will provide the opportunity for patients to enter a comprehensive medical history, from symptoms to lab results to medications and other treatment regimens.

This registry is entirely patient-driven; no medical records will be requested by the investigator, nor are visits with the investigator or any other research personnel required.

The registry database will be periodically "cleaned"; that is, records will be reviewed for duplication of entries and consistency of data. Many data validation checks are incorporated into the registry. Additional data clarification may be requested from users if users have chosen to provide an email address for contact.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* G1D diagnosis
* Patients experiencing symptoms of G1D but who have not yet received a diagnosis

Exclusion Criteria:

* Patients who are not experiencing any symptoms of G1D

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from the investigator's patients at the Rare Brain Disorders Clinic and from the national and international community of patients with Glucose Transporter Type I Deficiency
Sampling Method: Non-Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2013-12; Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Symptom Severity | 5 years
  It is hypothesized that symptom severity will correspond to the degree of biochemical dysfunction or mutation type (when available). A broad range of symptoms and severity ratings are collected both retrospectively and prospectively.

CONTACTS AND LOCATIONS:
Overall Officials: Juan M. Pascual, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Marin-Valencia I, Good LB, Ma Q, Malloy CR, Pascual JM. Heptanoate as a neural fuel: energetic and neurotransmitter precursors in normal and glucose transporter I-deficient (G1D) brain. J Cereb Blood Flow Metab. 2013 Feb;33(2):175-82. doi: 10.1038/jcbfm.2012.151. Epub 2012 Oct 17. PMID 23072752
- [Background] Marin-Valencia I, Good LB, Ma Q, Duarte J, Bottiglieri T, Sinton CM, Heilig CW, Pascual JM. Glut1 deficiency (G1D): epilepsy and metabolic dysfunction in a mouse model of the most common human phenotype. Neurobiol Dis. 2012 Oct;48(1):92-101. doi: 10.1016/j.nbd.2012.04.011. Epub 2012 Apr 23. PMID 22683290
- [Background] Marin-Valencia I, Roe CR, Pascual JM. Pyruvate carboxylase deficiency: mechanisms, mimics and anaplerosis. Mol Genet Metab. 2010 Sep;101(1):9-17. doi: 10.1016/j.ymgme.2010.05.004. Epub 2010 Jun 9. PMID 20598931
- [Background] Wang D, Sands T, Tang M, Monani U, De Vivo D. Glucose Transporter Type 1 Deficiency Syndrome. 2002 Jul 30 [updated 2025 Mar 6]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1430/ PMID 20301603
- [Background] Perez-Duenas B, Prior C, Ma Q, Fernandez-Alvarez E, Setoain X, Artuch R, Pascual JM. Childhood chorea with cerebral hypotrophy: a treatable GLUT1 energy failure syndrome. Arch Neurol. 2009 Nov;66(11):1410-4. doi: 10.1001/archneurol.2009.236. PMID 19901175
- [Background] Pascual JM, Campistol J, Gil-Nagel A. Epilepsy in inherited metabolic disorders. Neurologist. 2008 Nov;14(6 Suppl 1):S2-S14. doi: 10.1097/01.nrl.0000340787.30542.41. PMID 19225367
- [Background] Pascual JM, Wang D, Hinton V, Engelstad K, Saxena CM, Van Heertum RL, De Vivo DC. Brain glucose supply and the syndrome of infantile neuroglycopenia. Arch Neurol. 2007 Apr;64(4):507-13. doi: 10.1001/archneur.64.4.noc60165. Epub 2007 Feb 12. PMID 17296829
- [Background] Pascual JM, Wang D, Lecumberri B, Yang H, Mao X, Yang R, De Vivo DC. GLUT1 deficiency and other glucose transporter diseases. Eur J Endocrinol. 2004 May;150(5):627-33. doi: 10.1530/eje.0.1500627. PMID 15132717
- [Background] Pascual JM, Wang D, Yang R, Shi L, Yang H, De Vivo DC. Structural signatures and membrane helix 4 in GLUT1: inferences from human blood-brain glucose transport mutants. J Biol Chem. 2008 Jun 13;283(24):16732-42. doi: 10.1074/jbc.M801403200. Epub 2008 Apr 3. PMID 18387950
- [Background] Pascual JM. [Glucose transport hereditary diseases]. Med Clin (Barc). 2006 Nov 11;127(18):709-14. doi: 10.1157/13095099. Spanish. PMID 17169300
- [Background] Wang D, Pascual JM, Yang H, Engelstad K, Mao X, Cheng J, Yoo J, Noebels JL, De Vivo DC. A mouse model for Glut-1 haploinsufficiency. Hum Mol Genet. 2006 Apr 1;15(7):1169-79. doi: 10.1093/hmg/ddl032. Epub 2006 Feb 23. PMID 16497725
- [Background] Wang D, Pascual JM, Yang H, Engelstad K, Jhung S, Sun RP, De Vivo DC. Glut-1 deficiency syndrome: clinical, genetic, and therapeutic aspects. Ann Neurol. 2005 Jan;57(1):111-8. doi: 10.1002/ana.20331. PMID 15622525
- [Background] Pascual JM, Lecumberri B, Wang D, Yang R, Engelstad K, De Vivo DC. [Type 1 glucose transporter (Glut1) deficiency: manifestations of a hereditary neurological syndrome]. Rev Neurol. 2004 May 1-15;38(9):860-4. Spanish. PMID 15152356
- [Background] Wang D, Pascual JM, Iserovich P, Yang H, Ma L, Kuang K, Zuniga FA, Sun RP, Swaroop KM, Fischbarg J, De Vivo DC. Functional studies of threonine 310 mutations in Glut1: T310I is pathogenic, causing Glut1 deficiency. J Biol Chem. 2003 Dec 5;278(49):49015-21. doi: 10.1074/jbc.M308765200. Epub 2003 Sep 16. PMID 13129919
- [Background] Pascual JM, Van Heertum RL, Wang D, Engelstad K, De Vivo DC. Imaging the metabolic footprint of Glut1 deficiency on the brain. Ann Neurol. 2002 Oct;52(4):458-64. doi: 10.1002/ana.10311. PMID 12325075
- [Background] Iserovich P, Wang D, Ma L, Yang H, Zuniga FA, Pascual JM, Kuang K, De Vivo DC, Fischbarg J. Changes in glucose transport and water permeability resulting from the T310I pathogenic mutation in Glut1 are consistent with two transport channels per monomer. J Biol Chem. 2002 Aug 23;277(34):30991-7. doi: 10.1074/jbc.M202763200. Epub 2002 May 24. PMID 12032147
- [Background] De Vivo DC, Wang D, Pascual JM, Ho YY. Glucose transporter protein syndromes. Int Rev Neurobiol. 2002;51:259-88. doi: 10.1016/s0074-7742(02)51008-4. No abstract available. PMID 12420362
- [Background] Brockmann K, Wang D, Korenke CG, von Moers A, Ho YY, Pascual JM, Kuang K, Yang H, Ma L, Kranz-Eble P, Fischbarg J, Hanefeld F, De Vivo DC. Autosomal dominant glut-1 deficiency syndrome and familial epilepsy. Ann Neurol. 2001 Oct;50(4):476-85. doi: 10.1002/ana.1222. PMID 11603379